CLINICAL TRIAL: NCT01350089
Title: A Double Blind, Randomised, Placebo-controlled, Within-subject Crossover Study to Examine the Possible Effects of Energy Drink Ingestion on Perceived Alcohol Intoxication
Brief Title: Possible Effects of Energy Drink Ingestion on Perceived Alcohol Intoxication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Univ. Prof. Dr. Christoph Aufricht, Medical University of Vienna, Department of Pediatrics and Adolescent Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ED and alcohol intoxication
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Perceived Alcohol Intoxication
Keywords: energy drinks; alcohol intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Ethanol; Caffeine; Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (without alcohol, caffeine, energy drink)
- Comparator 1 (with alcohol) (Active Comparator)
  Interventions: Drug: Comparator 1 (with alcohol; without caffeine and energy drink)
- Comparator 2 (with alcohol and coffeine) (Active Comparator)
  Interventions: Drug: Comparator 2 (with alcohol and caffeine; without energy drink)
- Comparator 3 (with alcohol and energy drink) (Experimental)
  Interventions: Drug: Comparator 3 (with alcohol and energy drink)

INTERVENTIONS:
Drug: Placebo (without alcohol, caffeine, energy drink) — (carbonated) water (volume equivalent to 46.5 g ethanol (inform of vodka (37.5%)) (carbonated) water (250 ml), artificial fruit juice (21 g/L prepared with (carbonated) water). The final volume of the mixture is 500 mL.
  Arms: Placebo
Drug: Comparator 1 (with alcohol; without caffeine and energy drink) — Mixture of 46.5 g ethanol (inform of vodka (37.5%)), (carbonated) water 250 mL, artificial fruit juice (21 g/L prepared with (carbonated) water). The final volume of the mixture 500 mL.
  Arms: Comparator 1 (with alcohol)
Drug: Comparator 2 (with alcohol and caffeine; without energy drink) — Mixture of 46.5 g ethanol (inform of vodka (37.5%)), caffeine (80 mg), (carbonated) water (250 ml), artificial fruit juice (21 g/L prepared with (carbonated) water) The final volume of the mixture is 500 mL.
  Arms: Comparator 2 (with alcohol and coffeine)
Drug: Comparator 3 (with alcohol and energy drink) — Mixture of 46.5 g ethanol (inform of vodka (37.5%)), Red Bull® Energy Drink (250 mL, without flavour mixture to optimize blinding), artificial fruit juice (21 g/L prepared with (carbonated) water).The final volume of the mixture is 500 mL.
  Arms: Comparator 3 (with alcohol and energy drink)

SUMMARY:
The purpose of this study is to determine whether the ingestion of caffeine, Energy Drinks has an effect on perceived alcohol intoxication.

DETAILED DESCRIPTION:
In each of the four study periods, subjects will receive one of the four study treatments in a double blind, randomised, manner. The effects of study treatment on alcohol intoxication will be determined by measurement of breath alcohol concentration and subjective effects of intoxication. Safety and tolerability will be monitored by measurement of vital signs, in particular pulse, and review of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Able and willing to comply with the requirements of the study, confirmed by written informed consent
* Aged 20 to 26 years
* Within acceptable range for weight and body mass index (70-85 kg and 21 to 25 kg/m2)
* At least 12-14 years of formal education
* In good general health as determined by medical history and screening investigations (see below)
* Taking no regular medication
* No history of psychiatric disorders
* Moderate alcohol consumption (less than 190.4 g/week) according to the Daily Drink questionnaire (Collins et a., 1985)
* "sporadic" users of Energy Drinks (fewer than 10 cans of 250 ml in the last 6 months)
* Confirmation that the general practitioner/primary care physician knows no reason that would prevent their participation
* Similar in social and demographic data, similar quality of life
* similar patterns of use of alcoholic beverages and Energy Drinks as well as quality of life (Martinez et al., 2000)
* similar level of physical activity (physical activity questionnaire) (Baecke et al., 1982)

Exclusion Criteria:

* Any condition that the investigator and/or sponsor consider might increase the risk to the volunteer or decrease the chance of obtaining satisfactory data
* Consumed 2>x>4 caffeine-containing drinks/day within 3 months of screening
* Smoked >10 cigarettes/day or equivalent within 3 months of screening
* Consumed more than 190.4 g alcohol per week, or have a history of alcohol or drug abuse or
* Consumed less than one alcoholic drink per week

Ages: 20 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Changes in breath alcohol concentration | from baseline up to 150 minutes
Changes of subjective effects of intoxication | from baseline up to 120 minutes

SECONDARY OUTCOMES:
Safety and tolerability | participants will be followed for the whole testing period of an expected average of 5 hours
  Safety and tolerability will be monitored by measurement of vital signs, in particular pulse, and review of adverse events.
Changes in Supine and standing vital signs | from baseline up to 150 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Aufricht, Univ.Prof.Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Deparment of pediatric and adolescent medicine, Vienna, Austria

REFERENCES:
- See also: Homepage MUVienna — http://www.meduniwien.ac.at